CLINICAL TRIAL: NCT04476147
Title: The Impact of Frailty on Thrombosis of Elderly Patients With Non-valvular Atrial Fibrillation (NVAF).
Brief Title: The Impact of Frailty on Thrombosis of Elderly Patients With NVAF （FTE-NVAF）
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hongwei Li, MD, Prof., Beijing Friendship Hospital
Other Study IDs: BFH - Frailty and thrombosis
Record Dates: First submitted 2020-07-15; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Non-valvular Atrial Fibrillation, Elderly, Frailty, Thrombosis
MeSH Terms: conditions — Frailty; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participates: This is an observational study
  Interventions: Other: Diagnostic Test: CHA2DS2-VASc, HAS-BLED and Fried Scale.

INTERVENTIONS:
Other: Diagnostic Test: CHA2DS2-VASc, HAS-BLED and Fried Scale. — This is an observational study. All the patients evaluate with CHA2DS2-VASc, HAS-BLED and Fried Scale, and observe the incidence of thrombotic events and the influence of frailty on thrombotic events in elderly patients with NVAF.

SUMMARY:
This study aims to investigate the use of anticoagulants in elderly patients with non-valvular atrial fibrillation (NVAF) and the incidence of frailty in elderly patients with NVAF. After two years follow-up, we observe the incidence of thrombotic events and the influence of frailty on thrombotic events in elderly patients with NVAF.

ELIGIBILITY:
Inclusion Criteria:

* ≥65yr
* Confirmed non-valvular atrial fibrillation (NVAF) diagnosis with ECG or Holter
* fulfilled CHA2DS2-VASc, HAS-BLED and Fried Scale
* patients agreed and provided informed consent

Exclusion Criteria:

* valvular atrial fibrillation
* cardiac surgery related atrial fibrillation
* acute disease related atrial fibrillation
* patients not fulfilled all the exam and text，or not accept the follow-up

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The inhospital patients (≥65yr) with NVAF of Beijing Friendship Hospital, Capital Medical University
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Ischemic stroke | 24 months
  Cerebral infarction, Transient ischemic attack, Cerebral embolism.
Massive hemorrhage | 24 months
  Life-threatening or imminently fatal bleeding, intracranial, retroperitoneal, compartment syndrome, massive gastrointestinal, etc.
All-cause death | 24 months
  All-cause death during the 2-year observation

CONTACTS AND LOCATIONS:
Overall Officials: Yunli Xing, Dr., Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Background] Xing Y, Ma Q, Ma X, Wang C, Zhang D, Sun Y. CHADS2 score has a better predictive value than CHA2DS2-VASc score in elderly patients with atrial fibrillation. Clin Interv Aging. 2016 Jul 14;11:941-6. doi: 10.2147/CIA.S105360. eCollection 2016. PMID 27478371
- [Background] Xing YL, Ma Q, Ma XY, Wang CY, Zhou Z, Huang YS, Sun Y. Characteristics of non-valvular atrial fibrillation patients who benefit most from anticoagulation treatment. Int J Clin Exp Med. 2015 Oct 15;8(10):18721-8. eCollection 2015. PMID 26770487
- [Background] Fumagalli S, Said SAM, Laroche C, Gabbai D, Marchionni N, Boriani G, Maggioni AP, Popescu MI, Rasmussen LH, Crijns HJGM, Lip GYH; EORP-AF Investigators. Age-Related Differences in Presentation, Treatment, and Outcome of Patients With Atrial Fibrillation in Europe: The EORP-AF General Pilot Registry (EURObservational Research Programme-Atrial Fibrillation). JACC Clin Electrophysiol. 2015 Aug;1(4):326-334. doi: 10.1016/j.jacep.2015.02.019. Epub 2015 Apr 20. PMID 29759321
- [Background] Bo M, Li Puma F, Badinella Martini M, Falcone Y, Iacovino M, Grisoglio E, Bonetto M, Isaia G, Ciccone G, Isaia GC, Gaita F. Health status, geriatric syndromes and prescription of oral anticoagulant therapy in elderly medical in-patients with atrial fibrillation: a prospective observational study. Int J Cardiol. 2015;187:123-5. doi: 10.1016/j.ijcard.2015.03.334. Epub 2015 Mar 21. No abstract available. PMID 25828331
- [Background] Mazzone A, Bo M, Lucenti A, Galimberti S, Bellelli G, Annoni G. The role of comprehensive geriatric assessment and functional status in evaluating the patterns of antithrombotic use among older people with atrial fibrillation. Arch Gerontol Geriatr. 2016 Jul-Aug;65:248-54. doi: 10.1016/j.archger.2016.04.008. Epub 2016 Apr 13. PMID 27131228